CLINICAL TRIAL: NCT05858996
Title: Testing the Pain Clinical Practice Guideline Using the Evidence Integration Triangle
Brief Title: Testing the Pain Clinical Practice Guideline
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Barbara Resnick, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00105286
Record Dates: First submitted 2023-04-25; First posted 2023-05-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pain; Dementia
MeSH Terms: conditions — Pain; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain-CPG-EIT (Experimental): The four components of the PAIN-CPG-EIT are provided by a research nurse facilitator working with the champion(s) and stakeholder team. Following the first stakeholder team meeting, the research nurse facilitator works 8 hours weekly during months one and two and then for four hours weekly months three to 12 to implement: Component I: Stakeholder team meeting and goal setting; Component II: Education of the staff; Component III: Mentoring and motivating the staff to address pain using the Pain Management CPG ; and Component IV: Ongoing monitoring of pain management in the community based on the Pain Management CPG.
  Interventions: Behavioral: Pain-CPG-EIT
- Pain-CPG-Education Only (Active Comparator): Communities randomized to education only will be provided with staff education using our developed Powerpoint for Component II of the PAIN-CPG-EIT intervention in 30 minute sessions as is currently done in usual practice. They will also be given access to an online copy of the Pain Management CPG. The education will be provided in the preferred format (e.g., face-to-face; webinar).
  Interventions: Other: Pain-CPG-Education Only

INTERVENTIONS:
Behavioral: Pain-CPG-EIT — Following randomization champions and stakeholder team members from the communities will be identified. The investigators will recommend the following individuals to be members of the stakeholder team: a nurse in a leadership position (e.g., director of nursing); the designated champion(s); nursing home administrator; physician/medical director, nurse practitioner and/or physician assistant; unit nurse; nursing assistant; activity staff; social worker; pharmacist; and rehabilitation therapists.
  Following the first stakeholder team meeting, treatment communities will be provided with a research nurse facilitator to work 8 hours weekly during months one and two and then for four hours weekly starting in month three for a total of 12 months to provide the four components of the PAIN-CPG-EIT.
  Arms: Pain-CPG-EIT
Other: Pain-CPG-Education Only — The Pain-CPG-Education only group will be provided with the same education as used in Component II of the Pain-CPG-EIT intervention. The education will be provided based on the preferences of the community (this may be face-to-face; online; or via handouts).
  Other Names: EO
  Arms: Pain-CPG-Education Only

SUMMARY:
There are evidence based processes for assessment and management of pain using pharmacologic and nonpharmacological approaches. These were reviewed and included within the Pain Management Clinical Practice Guideline (Pain Management CPG) recently developed by AMDA: The Society for Post-Acute and Long-Term Care Medicine. There are, however, many challenges to translating the use of Clinical Practice Guidelines into clinical settings. To overcome these challenges we developed and previously tested a theoretically based approach and merged this approach with the Pain Management CPG, which is referred to as the PAIN-CLINICAL PRACTICE GUIDELINE-USING THE EVIDENCE INTEGRATION TRIANGLE (PAIN-CPG-EIT). The PAIN-CPG-EIT involves a research nurse facilitator working with an identified community champion(s) and stakeholder team for 12 months to provide the following four components: Component I: Establishing and meeting monthly with a Stakeholder Team; Component II: Education of the staff; Component III: Mentoring and motivating the staff to address pain; Component IV: Ongoing evaluation of resident pain outcomes. Twelve communities will be included with 25 residents living with dementia and pain recruited from each community. Six communities will be randomized to treatment (PAIN-CPG-EIT) and six randomized to education only (EO) which involves providing the same education to staff as is done in Component II of PAIN-CPG-EIT. The primary aim of this study is to test the effectiveness of use of the PAIN-CPG-EIT to improve the assessment, diagnosis and management of pain and decrease pain intensity among nursing home residents living with dementia between baseline, 4 and 12 months and evaluate treatment fidelity. A secondary aim of the study is to consider differences in measurement, treatment and response to treatment between male and female and Black versus White residents living with dementia. Findings from this study will help build on the currently limited information about pain presentation and management among older adults living with dementia in nursing homes and improve health equity of aging populations experiencing pain.

DETAILED DESCRIPTION:
Pain is a common symptom among older adults in nursing home settings affecting 30% to 80% of residents living with dementia. Pain is not assessed, the underlying cause is not identified and treatment is not initiated for a large percentage of residents living with dementia in nursing homes. Lack of accurate pain evaluation results in untreated or over-treated pain. Untreated or over-treated pain can lower quality of life, negatively impact function, impair sleep, and increase behavioral and psychological symptoms associated with dementia. Reasons for lack of pain assessment, diagnosis and management for residents living with dementia include lack of knowledge among staff on how to evaluate and treat pain, limited options for complete pain relief, concerns related to use of opioids, and beliefs that pain is a normal part of aging among others.

For those with moderate to severe dementia verbal reporting of pain may not be reliable and observational approaches are recommended. Pain in individuals living with dementia is more likely to present with aggression, agitation, repetitive vocalizations, restlessness, sleep disturbances, withdrawal, and apathy and may be incorrectly treated with psychotropic medications. Evaluation and management of pain is also complicated by differences between sex/gender, racial and ethnic groups. In some studies individuals living with dementia who were older, male, or Black were less likely to verbally report having pain or to be treated for pain compared to those who were younger, female, or white. With regard to treatment, there is some evidence that nonpharmacological treatments and analgesics can decrease pain among individuals living with dementia. Engaging individuals, particularly those living with dementia, in interventions to manage pain such as physical activity or positioning can be difficult and staff need education and techniques to use to motivate residents in these activities.

Evidence based pain assessment, diagnosis and management approaches for nursing home residents, including residents living with dementia, were recently incorporated into a new Pain Management Clinical Practice Guideline (Pain CPG). Translation of Clinical Practice Guidelines or evidence based practices into real world settings are slow to occur and innovative approaches are needed. In prior work to facilitate translation of best practices the investigators developed a successful theoretically based approach that utilized the Social Ecological Model and Social Cognitive Theory and was guided by the Evidence Integration Triangle. Using this theoretically based approach there was a change in staff and resident behavior related to increasing residents' physical activity using a function focused care approach and increased use of nonpharmacological approaches to address behavioral symptoms associated with dementia. The purpose of this study is to utilize the previously established theoretically based approach to translate use of the new Pain Management CPG into nursing home settings and improve the assessment, diagnosis and management of pain among residents living with dementia. The theoretically based approach combined with the Pain Management CPG is referred to as the PAIN-CPG-EIT. The PAIN-CPG-EIT is initiated by a research nurse facilitator who works with community champions and a stakeholder team for 12 months to provide four components: Component I: Establishing and meeting monthly with a stakeholder team and champion(s) to establish community goals related to pain and review the Pain Management CPG; Component II: Education of the staff about assessment, diagnosis and management of pain of residents living with dementia based on the Pain Management CPG; Component III: Mentoring and motivating staff to assess, diagnose and manage pain; and Component IV: Ongoing monitoring of pain assessment, diagnosis and management and feedback to the stakeholder team. Twelve communities will be randomized to treatment (PAIN-CPG-EIT) or Education Only (EO) and 25 residents living with dementia and pain will be recruited per community. The first aim of this study is to: Test the effectiveness of use of the PAIN-CPG-EIT to improve the assessment, diagnosis and management of pain and decrease pain intensity among nursing home residents living with dementia. The second aim is to evaluate treatment fidelity related to use of the PAIN-CPG-EIT based on delivery, receipt and enactment. The third aim is to: a. test for gender/sex and race invariance in pain measurement based on the Pain in Alzheimer's Disease (PAIN-AD) measure; and b. test for differences in treatment of pain and response to treatment between male and female and Black versus White residents living with dementia. Findings will help to improve the assessment, diagnosis and management of pain and evaluate health disparities and equity among older adults living with dementia experiencing pain. Demonstrating effectiveness of this approach to using the Pain Management CPG will facilitate future work disseminating and implementing this CPG.

ELIGIBILITY:
Inclusion Criteria:

* Living in a participating community
* 60 years of age or older
* Evidence of dementia based on a score of 0-12 on the Brief Interview of Mental Status (BIMS); a score of >2 on the AD8 Dementia Screening Interview; a score of 0.5 to 2.0 on the Clinical Dementia Rating Scale (CDR); and lastly to differentiate between dementia and mild cognitive impairment a score of 9 or greater on the Functional Activities Questionnaire (FAQ).
* have evidence of pain at the time of recruitment based on the Minimum Data set assessment item: How much of the time over the past 5 days have you experienced pain or hurting with eligibility based on the following responses or evidence: occasionally, frequently or almost constantly, or staff report of pain at the same frequency; or if the resident is receiving nonpharmacological or pharmacological treatment for pain.

Exclusion Criteria:

* admitted to the nursing home for short-stay rehabilitation or other subacute needs (e.g., intravenous antibiotics);
* receiving Hospice care.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
pain assessment completed | baseline
  whether or not an appropriate pain assessment is completed
pain assessment completed | four months
  whether or not an appropriate pain assessment is completed
pain assessment completed | twelve months
  whether or not an appropriate pain assessment is completed
Pain management in careplan | baseline
  evidence that there is a pain management plan in the careplan
Pain management in careplan | 4 months
  evidence that there is a pain management plan in the careplan
Pain management in careplan | 12 months
  evidence that there is a pain management plan in the careplan
Appropriate use of opioids | baseline
  Review of 10 factors that indicate that opioids are being used appropriately as per the CPG. scores can range from 0 to 10 and higher scores indicate more appropriate use of opioids.
Appropriate use of opioids | four months
  Review of 10 factors that indicate that opioids are being used appropriately as per the CPG. scores can range from 0 to 10 and higher scores indicate more appropriate use of opioids.
Appropriate use of opioids | 12 months
  Review of 10 factors that indicate that opioids are being used appropriately as per the CPG. scores can range from 0 to 10 and higher scores indicate more appropriate use of opioids.

SECONDARY OUTCOMES:
Pain in Alzheimer's Disease (PAIN-AD) | baseline
  The PAIN-AD is a 5 item observation measure of pain for older adults living with dementia. Scores can range from 0 to 10 and higher scores indicate more pain
Pain in Alzheimer's Disease (PAIN-AD) | 4 months
  The PAIN-AD is a 5 item observation measure of pain for older adults living with dementia. Scores can range from 0 to 10 and higher scores indicate more pain.
Pain in Alzheimer's Disease (PAIN-AD) | 12 months
  The PAIN-AD is a 5 item observation measure of pain for older adults living with dementia. Scores can range from 0 to 10 and higher scores indicate more pain.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Future Care Coldspring, Baltimore, Maryland
  - Future Care Courtland, Baltimore, Maryland
  - Futurecare Northpoint, Baltimore, Maryland
  - Futurecare Irvington, Baltimore, Maryland
  - Communicare Ellicott City, Ellicott City, Maryland
  - communicare Marley Station, Glen Burnie, Maryland
  - Charles E Smilth Life Community, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: Yes
The plan is to provide any information requested by other researchers with a plan for rationale for the request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study and following publication of major outcome paper.
Access Criteria: Request from others